CLINICAL TRIAL: NCT01006421
Title: Oral Ginkgo Biloba and Narrow Band UVB in the Treatment of Vitiligo : A Randomized Double - Blind Placebo Controlled Trial
Brief Title: Oral Ginkgo Biloba and Narrow Band UVB in the Treatment of Vitiligo
Acronym: GB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Collaborators: University Hospital (Other)
Responsible Party: DR KHALID ALGHAMDI, KSU
Other Study IDs: GB-NBVUB
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Vitiligo
Keywords: phototherapy; Gingko biloba; repigmentation
MeSH Terms: conditions — Vitiligo | interventions — Ginkgo Extract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: GINGKO BILOBA — MEMOREX 60 MG BID

SUMMARY:
Vitiligo is a common chronic skin disease with 1-4% prevalence. It has a significant psychosocial impact on patients and society. Different treatment modalities with variable success rates are available.

Phototherapy is among the successful treatments but gives modest results. Some reports documented the usefulness of Ginkgo Biloba (GB) when used alone in Vitiligo treatment.

DETAILED DESCRIPTION:
Adding GB to phototherapy, especially the most commonly used one; Narrow-Band UVB (NBUVB) might give better results than using either one alone. This might improve repigmentation as well as patients' quality-of-life. (QOL).

This will be a prospective double-blind randomized controlled clinical trial. One-hundred-sixty Vitiligo patients will be randomly divided into 2 groups( 80 patients per group).

One group will receive oral GB (2 tablets of 60 mgs twice daily) with NBUVB twice weekly.

The other group will receive placebo tablets( identical in size, shape and color) to GB twice daily with NBUVB twice weekly.

Both groups will be treated for 6 months. Standard protocol of phototherapy will be used for both groups.

Our aim here is to see whether adding GB to NBUVB will lead to better repigmentation than placebo or not.

ELIGIBILITY:
Inclusion Criteria:

* Any Vitiligo patient (age 12 years and above) with non-segmental Vitiligo.
* Body surface area (BSA) involvement ≥ 3%.

Exclusion Criteria:

* Unable to consent
* Any topical, systemic or phototherapy for Vitiligo in the previous 2 months.
* Pregnancy, breast feeding.
* Liver or kidney disease.
* Epilepsy
* Bleeding disorder or anticoagulant treatment

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DERMATOLOGY CLINIC
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-01; Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Repigmentation (more than 50% from baseline) as the primary outcome | 3,6 and 9 months

SECONDARY OUTCOMES:
Quality-of-life - as secondary outcome . | 3,6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: KHALID M ALGHAMDI, MD, Study Chair — KSU
Locations (1):
- King Khalid University Hospital, Riyadh, Central, Saudi Arabia